CLINICAL TRIAL: NCT04287192
Title: Digital Bridge: Using Technology to Support Patient-centered Care Transitions From Hospital to Home
Acronym: DB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); Trillium Health Partners (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Digital Bridge
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-11

CONDITIONS: Older Adults With Complex Care Needs

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a non-randomized control trial to understand the impact of the intervention. For each site (Sinai Health System and THP - both Mississauga and Credit Valley sites) and each service, half of the participating wards will be designated as control while the other half will be designated as intervention. The investigators will collect baseline data from all wards (control and intervention) during phase 1 while co-design is on-going and the intervention has not been deployed. During phase 2, after co-design is complete, the co-designed technology intervention and workflow will be rolled out to only the intervention wards. The investigators will then collect data (identical to what was collected at baseline) from all wards (control and intervention) to understand the impact of technology by examining the differential change between control and intervention wards (difference in difference approach).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Control: Control participants will complete surveys at 4 time points (baseline, 1-2 weeks, 3 month and 6 months after discharge). The surveys will capture data on demographics, assess their transition quality, self-reported costs, and assess their quality of life. Aside from completion of these surveys, no changes to their usual care will occur.
- (Digital Bridge intervention) (Experimental): Experimental (Digital Bridge intervention) participants will complete surveys at 4 time points (baseline, 1-2 weeks, 3 month and 6 months after discharge). The surveys will capture data on demographics, assess their transition quality, self-reported costs, assess their quality of life, and goal attainment.
  One to two days before discharge, patients will work with their team to develop the PODS in Care Connector. Once the PODS is created, the patient and hospital provider will be prompted to set transition goals using the ePRO tool.
  Interventions: Other: Digital Bridge:Tool Intervention

INTERVENTIONS:
Other: Digital Bridge:Tool Intervention — Our Digital Bridge is an integration of the Care Connector and ePRO technologies that will support care transitions by: 1) inviting PCPs to access Care Connector while the patient is in hospital, allowing for asynchronous communication via the messaging feature for proactive discharge planning, 2) facilitating the inclusion of inter-professional recommendations in the discharge module (e.g. diet and mobility) typically missing from traditional physician generated discharge summaries, 3) electronic generation of PODS for use in patient-centred discharge teaching, 4) providing patients electronic access to PODS post discharge to facilitate use of information at home, 5) adoption of digital enabled goal-oriented process to engage patients and families in discharge process, and 6) providing ongoing self-management support for patients using ePRO for the vulnerable period 6 months post discharge.
  Arms: (Digital Bridge intervention)

SUMMARY:
Older adults who live with multiple chronic conditions are more likely to experience frequent admissions and discharges from hospital. These transitions are often challenging and leave people at risk of readmission. Appropriate, timely and person-centred communication across all health care providers involved in transitions (in and out of hospital) as well as with patients and their families is critical to ensure a smooth and effective transition process. Digital health technologies can play an important role in improving person-centred communication across clinical settings and clinicians. This project will develop and test a Digital Bridge by connecting communication technologies already in use in hospital and primary care/community settings to improve communication between providers in hospital and in primary care, patients and family caregivers from admission to 6 months post-discharge. The investigators will engage with all the technology users to co-design the Digital Bridge, ensuring that how the investigators connect the existing technologies and adopt them into practice will meet the needs of providers, patients and their caregivers. Next hospital partners will adopt the technology into general medicine and rehabilitation services in hospital systems in Toronto (Sinai Health System) and Mississauga (Trillium Health Partners). The investigators will evaluate the Digital Bridge through a pre-post pragmatic trial, assessing impact on patient experience (quality of transition), patient outcomes (quality of life), transition processes (provider communication and teamwork), and system costs (economic evaluation). This project adopts an implementation science lens, allowing the investigators to collect qualitative data on enablers and barriers to adopting the Digital Bridge to help inform development of a scale and spread strategy.

DETAILED DESCRIPTION:
Older adults with multi-morbidity and complex care needs (CCN) are among those most likely to experience frequent care transitions between settings, particularly from hospital to home. Many of these community-dwelling older adults fall into the category of high-cost users, who account for the majority of year over year healthcare spending in Ontario, Canada and internationally. The complexity of these individuals stems not only from their multimorbidity disease profiles, but also the social, environmental and contextual issues that make it difficult for them to manage their physical health needs. It is often the interaction of these challenges which results in frequent visits to the hospital.

When patients leave the hospital, they face challenges as they attempt to cope and adjust at home. Krumholz coined the term 'post-hospital syndrome' to describe this acquired, transient period of vulnerability post-discharge due to impaired physiological systems and depleted reserves. This depletion limits patients' ability to adjust and manage their health issues, often leading to hospital re-admission within 30 days with an acute medical illness unrelated to the original diagnosis. Poor communication and incomplete information transfer between the various clinicians and organizations providing care to CCN patients as they transition from hospital to home can impede access to needed support and resources during this vulnerable time. Studies have demonstrated that insufficient communication during the transition process can lead to poor patient outcomes and higher rates of readmission for older adults with CCN.

While improving clinician communication is important, the quality and content of that communication with patients also matters. Patients with CCN benefit most from person-centred delivery models that can adapt to their unique needs and engage them as partners in their care. Person-centred approaches have been shown to improve discharge from hospital to home by emphasizing partnership between patient and provider, improving patient self-efficacy, and through improving communication between patients, providers and within care teams. For patients with CCN, incorporating ongoing support for self-care after they return home as part of that communication can offer additional support and benefit. In sum, communication that enables person-centred care and supported self-management may offer the greatest advantages as the investigators support older adults with complex care needs transitioning from hospital to home.

Digital health technologies offer a promising and appealing solution to support this type of person-centred communication across inter-professional teams working within and between health care organizations. A systematic review of inter-professional communication in transitional care models found that information systems, as well as multi-professional care coordination support higher satisfaction and subjective quality of life for older adults. A key strength of digital solutions is their ability to foster shared situational awareness of inter-professional teams. An essential component of interdisciplinary communication, shared situational awareness is a group or team's ability to understand the "big picture" and work together towards a common goal, like transitioning a patient from hospital to home.

While these examples demonstrate the potential of digital communication platforms to improve team communication and functioning, there remain a number of issues that limit the value of current systems. First, the majority of communication systems exist within single teams or organizations, and rarely span those boundaries. Second, many available communication systems do not inherently support person-centred care delivery, as few are co-designed with patients and providers. As such, many of the available systems are not well suited to supporting the communication needs of care teams, patients and families during the time of transition from hospital back to the community. Finally, many existing systems have only been evaluated over short-periods with insufficient attention to implementation as a means to support both evidence of effectiveness as well as transferability of findings.

This project will address these three gaps by implementing and evaluating a Digital Bridge to support person-centred health care transitions for older adults with complex care needs. The Digital Bridge will: 1) span organizational and professional boundaries by enabling communication between inter-disciplinary teams working in hospital and primary care, with patients and caregivers; 2) support person-centred delivery through adoption of co-design methods to establish a workflow; and 3) be evaluated through an implementation science lens.

The Digital Bridge will integrate two tested and validated technologies that are currently in use in hospital and community settings: 1) Care Connector and 2) The electronic Patient Reported Outcomes (ePRO) tool. Care Connector is an inter-professional communication and collaboration platform initially designed in the hospital setting to support clinical teams caring for patients with CCN. The tool includes discharge communication supports like Patient Oriented Discharge Summaries (PODS), to support clinician communication and collaboration in the community and across care settings. The ePRO tool is a primary-care facing technology, co-designed with patients with CCN, their primary care providers and family caregivers to enable communication on patient-oriented goals. The investigators hypothesize that these two technologies will work synergistically by both supporting the communication and collaboration needs of clinicians and patients at the critical time of care transitions (Care Connector) and engaging patients to set goals and monitor their progress with clinicians starting in the hospital and through their transition back into the community over the longer term (ePRO).

ELIGIBILITY:
Inclusion Criteria:

* Patients with anticipated discharge home will be recruited at the time of admission to one of the services (i.e medicine or rehab) in the study. Patients aged 60 and over, with CCN defined as presenting with 3 or more chronic conditions from the 16 most prominent in the population, which is an established method to identifying patients with CCN. As the technology is only currently available in English, patients (or a caregiver) must be able to speak and read English. Patients with mild cognitive impairment will not be excluded if able to provide informed consent, and engage with the intervention (independently or with caregiver aid).

Exclusion Criteria:

* Previously participated in the study (in case of re-admission); discharge destination is another acute care facility, palliative care unit, complex continuing care, or long term care; died in hospital, cannot be contacted by telephone after discharge; unable to respond to survey question for any reason and lack of availability of family members and/or other caregivers willing and able to provide assistance.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Care Transitions Measure (CTM3) | At 1-2 weeks post-discharge
  The CTM3 is a patient-reported measure of transition quality focusing on person-centredness and communication; appropriate as the focus of the Digital Bridge is to improve person-centred communication during transitions. The CTM-3 survey has been validated in similar patient populations transitioning from hospital to home and primary care, and in a systematic review of transitions measures was deemed to be the most acceptable measure of quality transitions.

SECONDARY OUTCOMES:
Assessment for Quality of Life Scale 4D -AQoL-4D | At baseline, 1-2 weeks, 3 and 6 months post-discharge
  a brief survey validated in similar populations, with demonstrated responsiveness and predictive validity with regard to entrance to long-term care
Patient information sheet | Baseline
  This questionnaire will capture patient demographic and characteristic information such as age, gender, ethnicity, chronic illness profile, socio-economic status, and IT skills using the Patient Demographic forms.
Provider information sheet | Baseline
  This questionnaire will capture provider demographic and characteristic information such as age, gender, ethnicity, chronic illness profile, socio-economic status, and IT skills using the Provider Demographic forms.
Post-Study System Usability Questionnaire: PSSUQ | At 1-2weeks, 3 and 6 months post-discharge
  This questionnaire is designed to give an opportunity to talk about the reactions to the system that was used. These responses will help understand what aspects of the system that everyone is particularly concerned about, and the aspects everyone was satisfied with.
Patient/Caregiver self-reported costs | At 3 and 6 months post-discharge
  This questionnaire will ask about time and expenses relating to managing health conditions.
Caregiver information sheet | Baseline
  This questionnaire will allow us to understand who the caregivers are that participated in the study, and this will allow us to make sense of the data that will be collected during the working groups in a meaningful way.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Steele Gray, PhD, Principal Investigator — Sinai Health System; Terence Tang, MD, Principal Investigator — Trillium Health; Michelle Nelson, PhD, Principal Investigator — Sinai Health System
Locations (1):
- Sinai Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The reported data (which includes patient information at the aggregate level) will be disseminated widely via reports, conference presentations, peer reviewed journal articles and other standard modes of knowledge translation.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available through 2022-2024.
Access Criteria: Open access peer reviewed journal publication

REFERENCES:
- [Derived] Singh H, Armas A, Law S, Tang T, Steele Gray C, Cunningham HV, Thombs R, Ellen M, Sritharan J, Nie JX, Plett D, Jarach CM, Thavorn K, Nelson MLA. How digital health solutions align with the roles and functions that support hospital to home transitions for older adults: a rapid review study protocol. BMJ Open. 2021 Feb 25;11(2):e045596. doi: 10.1136/bmjopen-2020-045596. PMID 33632755
- [Derived] Steele Gray C, Tang T, Armas A, Backo-Shannon M, Harvey S, Kuluski K, Loganathan M, Nie JX, Petrie J, Ramsay T, Reid R, Thavorn K, Upshur R, Wodchis WP, Nelson M. Building a Digital Bridge to Support Patient-Centered Care Transitions From Hospital to Home for Older Adults With Complex Care Needs: Protocol for a Co-Design, Implementation, and Evaluation Study. JMIR Res Protoc. 2020 Nov 25;9(11):e20220. doi: 10.2196/20220. PMID 33237037